CLINICAL TRIAL: NCT01621087
Title: Dietary Linoleic Acid for Secondary Prevention of Coronary Heart Disease and Death in the Sydney Heart Study: a Randomized Controlled Dietary Trial
Brief Title: Dietary Linoleic Acid for Secondary Prevention of Coronary Heart Disease and Death in the Sydney Heart Study: an RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Chris Ramsden, Clinical Investigator, National Institutes of Health Clinical Center (CC)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIHCC-E5744
Record Dates: First submitted 2012-06-04; First posted 2012-06-18 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Safflower Oil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Safflower oil (Experimental)
  Interventions: Other: Safflower oil
- Control group (no diet instruction) (No Intervention)

INTERVENTIONS:
Other: Safflower oil — Liquid safflower oil and safflower oil polyunsaturated margarine
  Arms: Safflower oil

SUMMARY:
The substitution of polyunsaturated fatty acids (PUFA) for saturated fatty acids (SFA) is a cornerstone of worldwide dietary advice for coronary heart disease (CHD) risk reduction. However, clinical CHD benefits specific to the omega-6 PUFA linoleic acid (LA), and distinct from omega-3 PUFAs, have not been established. The Sydney Diet-Heart Study (SDHS; 1966-1973) was a randomized controlled secondary CHD prevention trial testing whether selectively increasing omega-6 LA from safflower oil in place of SFA reduced CHD and improved survival. A full analysis of mortality outcomes has not been published. The investigators recovered the original SDHS dataset, which included detailed longitudinal dietary, smoking and coded mortality data, permitting evaluation of smoking relapse rates, and all-cause, CVD and CHD mortality outcomes by nutrient intake and duration of diet exposure. Data recovery also permitted the first complete meta-analysis of LA intervention trials on mortality outcomes.

Objectives are (1) to evaluate whether increasing dietary linoleic acid alters CVD and CHD mortality, and (2) to assess whether changes in smoking relapse rates contribute to observed mortality differences.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of myocardial infarction, angina, or coronary insufficiency
* Willingness to attend Coronary Clinic in Sydney Australia on a regular basis

Ages: 30 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 458 (Actual)
Dates: Start 1966-02; Primary Completion 1973-06 (Actual)

PRIMARY OUTCOMES:
Death, all-cause | Up to 7 years

SECONDARY OUTCOMES:
Death due to cardiovascular disease | Up to 7 years
Death due to coronary heart disease | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Ramsden, MD, Principal Investigator — National Institutes of Health (NIH)
Locations (1):
- Prince Henry Hospital Coronary Clinic, Sydney, Australia

REFERENCES:
- [Result] Woodhill JM, Palmer AJ, Leelarthaepin B, McGilchrist C, Blacket RB. Low fat, low cholesterol diet in secondary prevention of coronary heart disease. Adv Exp Med Biol. 1978;109:317-30. doi: 10.1007/978-1-4684-0967-3_18. No abstract available. PMID 727035
- [Derived] Ramsden CE, Zamora D, Leelarthaepin B, Majchrzak-Hong SF, Faurot KR, Suchindran CM, Ringel A, Davis JM, Hibbeln JR. Use of dietary linoleic acid for secondary prevention of coronary heart disease and death: evaluation of recovered data from the Sydney Diet Heart Study and updated meta-analysis. BMJ. 2013 Feb 4;346:e8707. doi: 10.1136/bmj.e8707. PMID 23386268